CLINICAL TRIAL: NCT07027007
Title: Prospective Observational Analysis of Circulating Endocan Levels in Patients Presenting With Acute Diverticulitis
Acronym: DIVENDO
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Luca Ghirardelli, MD, IRCCS Ospedale San Raffaele
Other Study IDs: DIVENDO STUDY
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diverticulitis
Keywords: endocan; acute diverticolitis; diverticulitis classification
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with acute diverticulitis: Patients admitted to the emergency department with acute diverticulitis classified according to WSES statements.

SUMMARY:
Quantify the level of endocan in blood samples collected from patients with acute diverticulitis in the emergency department. Determine if endocan levels are correlated with the severity of diverticulitis according to the WSES classification. Assess whether patients requiring emergency surgical intervention have higher endocan values compared to others.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed informed consent
* Patients who are affected by acute diverticulitis after clinical evaluation and imaging (i.e. u.s. or CeCT)

Exclusion Criteria:

* Immunosuppressed patients
* Patients suffering chronic inflammatory diseases
* Patients with concomitant malignancy, cardiac, renal and haepatic failure
* History of major vascular surgery (aneurysmectomy)
* Pregnant women
* Patients participating in other studies that may interfere with the outcome of the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by acute diverticulitis in the emergency department
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Endocan serum level at admission | The serum of the patients enrolled inthe study will be collected within two hours from emergency room registation and tested for ENDOCAN
  To evaluate the correlation between blood concentration of endocan and severity of diverticulitis

SECONDARY OUTCOMES:
Predictive value of endocan in determining which patients need emergency surgery | Patients will undergo diverticulitis evaluations (per WSES criteria) within 3 hours of Emergency room admission and study enrollment
  Concentration of endocan in grade 3-4 WSES compared to grade1-2
Prognostic value of endocan in determining the risk of recurrent diveritculitis | From discharge after definitive tretament till 12 months follow-up
  Concentration of endocan in patient who develop a recurrence after 1 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department IRCCS San Raffaele, Milan, milano, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code